CLINICAL TRIAL: NCT02006030
Title: Randomized, Open Label, Phase 2 Trial of ADI PEG 20 Plus Concurrent Transarterial Chemoembolization (TACE) Versus TACE Alone in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Ph 2 Trial of ADI PEG 20 Plus Concurrent Transarterial Chemoembolization (TACE) Vs TACE Alone in Patients With Unresectable Hepatocellular Carcinoma
Acronym: TACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2013-003
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2016-09

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma; Liver Cancer; ADI; ADI-PEG 20
MeSH Terms: conditions — Liver Neoplasms | interventions — ADI PEG20; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADI-PEG 20 + TACE (Experimental): ADI-PEG 20 plus concurrent transarterial chemoembolization
  Interventions: Drug: ADI-PEG 20; Drug: Transarterial chemoembolization
- Transarterial chemoembolization (TACE) (Active Comparator): transarterial chemoembolization alone
  Interventions: Drug: Transarterial chemoembolization

INTERVENTIONS:
Drug: ADI-PEG 20
  Other Names: arginine deiminase formulated with polyethylene glycol
  Arms: ADI-PEG 20 + TACE
Drug: Transarterial chemoembolization
  Other Names: TACE

SUMMARY:
Certain cancers require the amino acid arginine. Arginine deiminase (ADI) is an enzyme from microbes that degrade arginine. ADI has been formulated with polyethylene glycol and has been used to treat patients that have cancers that require arginine. In this study, the investigators will evaluate the response rate, as determined by the revised International Working Group recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC confirmed clinically or histologically or cytologically. A clinical diagnosis of HCC, using the 2010 Guideline of the American Association for the Study of Liver Diseases requires the presence of hepatic tumor(s) with image findings (e.g. sonography, CT or MRI) compatible with HCC, and no evidence of other gastrointestinal tumors (Bruix [2011] - Guideline, 2010).
2. Solitary hepatic tumor <8 cm in diameter or multifocal disease as evidenced by CT or MRI scan. Tumor volume ≥50% of liver organ or infiltrating HCC should be excluded.
3. Not a candidate for surgical resection or ablation of the tumor.
4. The target lesion must not have been treated previously with local therapy, including TACE. Prior local therapy (radiofrequency ablation, percutaneous ethanol injection, cryoablation, or surgery) to nontarget lesions is acceptable.
5. The subject must have received no more than 2 TACE (n≤ 2) or the previous TACE was performed longer than 2 months before enrollment.
6. Local therapy must have been completed at least 4 weeks before baseline scan.
7. Measurable disease using mRECIST criteria (Appendix A) and RECIST1.1 (Appendix B) criteria. At least 1 measurable lesion must be present.
8. Barcelona Clinic Liver Cancer (BCLC) staging classification B (intermediate stage) (Appendix C).

Exclusion Criteria:

1. 1. Candidate for potential curative therapies (i.e., resection or transplantation).
2. Prior allograft transplantation including liver transplantation.
3. Significant cardiac disease (New York Heart Association Class III or IV; Appendix F).
4. Serious infection requiring treatment with systemically administered antibiotics.
5. Pregnancy or lactation.
6. Expected non-compliance.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situations that would limit compliance with study requirements.
8. Subjects who have had any anticancer treatment within 2 weeks prior to week 1 visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Determine time to tumor progression (TTP) | 2 years estimated - course of study

SECONDARY OUTCOMES:
Tumor response rates | 2 years estimated - course of study

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital Taipei, Taiwan
Locations (4):
- Taiwan (4):
  - CMUH, Taichung
  - National Taiwan University Hospital, Taipei
  - TP-VGH, Taipei
  - CGMH-LK, Taoyuan District